CLINICAL TRIAL: NCT05042752
Title: Impact of Clinical Ultrasound in Patients With Heart Failure Treated in Home Hospitalization (AHF-CU)
Brief Title: Impact of Clinical Ultrasound in Patients With Heart Failure Treated in Home Hospitalization
Acronym: AHF-CU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lara Palacios (Other)
Responsible Party: Sponsor-Investigator, Lara Palacios, Medical Doctor, Fundacion Miguel Servet
Organization: Fundacion Miguel Servet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-AHF-CU
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Acute Heart Failure (AHF)
Keywords: Acute heart failure; Ultrasound; Hospital at home; Readmision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention arm (No Intervention): Standard care of AHF on a patient admitted on a HAH unit consists in physical examination and basic complementary tests
- Experimental arm (Experimental): Clinical ultrasound on HAH admitted patient. Clinical handheld Ultrasound consists of inferior vena cava diameter measurement and lung ultrasound protocol in order to guided Diuretic Therapy
  Interventions: Procedure: CLINICAL ULTRASOUND

INTERVENTIONS:
Procedure: CLINICAL ULTRASOUND — The intervention group will receive the standard care of treatment in AHF and the performance of CU.
  Arms: Experimental arm

SUMMARY:
The purpose of this study is to assess whether clinical ultrasound (CU)-guided treatment in acute heart failure (AHF) is superior to the standard care (SC)-guided treatment. We would like to see if using a portable ultrasound to guide diuretic therapy for AHF patients will prevent hospital readmissions in the setting of hospitalization at home (HAH). This study will use a handheld ultrasound called IVIZ-Sonosite and aims to see whether changing diuretic therapy based on the performance of the ultrasound will result in the less hospitalizations for heart failure as compared to performing just SC-guided therapy.

DETAILED DESCRIPTION:
AHF remains a leading cause of death in industrialized countries. Despite advances in medical treatment, an estimated 250,000-300,000 AHF patients are hospitalized in the United States each year for symptoms caused by low cardiac output. Although the events that cause acute decompensation are multifactorial, the common pathway associated with decreased ventricular function are autonomic dysfunction and fluid retention. It has been previously suggested that an estimated 50%-66% of CHF hospitalizations may be preventable with improved monitoring of fluid volume status. In Spain, more than 10% of discharged patients are readmitted within 30 days. AHF is one of the most frequent reasons for readmission, mainly because of congestion-related symptoms. The size and shape of the inferior vena cava and the presence of B lines have proven to be effective to estimate volume overload and to guide diuretic treatment in AHF on a hospital setting. At the same time, technology is quickly evolving and new approaches for clinical care are arising.

The aim of this study is two compare SC-guided therapy vs CU-guided therapy in AHF patients admitted on a HAH. We designed an open label clinical trial, in which patients are randomized into two groups: "ultrasound group" who undergoes CU together with SC and "control group" who undergoes SC only. Diuretic treatment will be tailored according to the findings of the SC together with the CU or according to the findings of the SC respectively. A total of 140 patients will be recruited, 70 patients on each arm. The outcome variables are readmission for AHF and other causes, mortality for AHF and other causes, and the combined event of readmission for AHF and mortality for AHF at one month and two months. The CU protocol will include both lung ultrasound and inferior vena cava measurement and will be performed with an ultraportable device (IVIZ-Sonosite). Standard care will involve physical examination and basic complementary tests.

The way patients end up admitted to HAH are transferences from the emergency room, from the internal medicine ward, from the clinics and from primary care. During admission, daily visits are carried out by the nursing staff (except when clinical stability and no need to intravenous treatment infusions) and every two days by the medical team. Admission in the HAH is always voluntary and patients can decide to return to hospital during HAH stay. In the HAH unit, there is a 24-hour telephone service coordinated by a specialized nurse on call.

ELIGIBILITY:
Inclusion Criteria:

* AHA documented
* HAH admission
* Informed consent
* 2 or more CU on the intervention group being one the day of admission

Exclusion Criteria:

* Life expectancy below 6 months
* Active tumors
* Interstitial lung disease
* Respiratory distress
* Pulmonary concussion
* Inotropic drugs on admission
* Patients coming from intensive care unit
* Intolerance or allergy to diuretic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Readmission due to AHF | At 30 days and 60 days
  Admission on the internal medicine ward for more than 24 hours due to AHF after being discharge from the AHA unit. We do not consider admission in the emergency room due to AHF after being discharge from the AHA unit.
Mortality due to AHF | At 30 days and 60 days
  Death related to an AHF episode after being discharge from the AHA unit.

SECONDARY OUTCOMES:
Readmission due to a cause different to AHF. | At 30 days and 60 days
  Admission on the internal medicine ward for more than 24 hours after being discharge from the AHA unit due to a cause different to AHF. We do not consider admission in the emergency room after being discharge from the AHA unit due to a cause different to AHF
Mortality due to a cause different to AHF | At 30 days and 60 days.
  Any death related to a cause different to AHF after being discharge from the AHA unit.

OTHER OUTCOMES:
Cumulative event | At one or two months
  At least one AHA readmission or mortality due to AHA

CONTACTS AND LOCATIONS:
Overall Officials: LARA PALACIOS GARCIA, MD, Principal Investigator — Hospital Reina Sofia
Locations (1):
- Hospital Reina Sofia, Tudela, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No